CLINICAL TRIAL: NCT04242914
Title: The Effect of Intravenous Ketamine on Non-suicidal Self-injuries in Women Suffering From Complex Post Traumatic Stress Disorder (cPTSD)
Brief Title: The Effect of Intravenous Ketamine on Non Suicidal Self Injuries.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0724-018-TLV
Record Dates: First submitted 2020-01-09; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Non Suicidal Self Injury
Keywords: Ketamine, Midazolam, Non-Suicidal Self-Injury, Intravenous
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: randomized control, double blind trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded participants and investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Research: Ketamine + Midazolam (Experimental): Research group will receive ketamine and midazolam.
  Interventions: Drug: Ketamine; Drug: Midazolam
- Control: Midazolam (Experimental): Control group will receive midazolam.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Intravenous Ketamine, dose 0.5mg/kg in 100ml Sodium Chloride 0.9% over 40 minutes.
  Arms: Research: Ketamine + Midazolam
Drug: Midazolam — Intravenous Midazolam, dose 0.03mg/kg in 100ml Sodium Chloride 0.9% over 40 minutes.

SUMMARY:
Non-suicidal self-injuries (NSSI) is a deliberate harm a person causes directly to their body, resulting in structural or functional damage, without suicidal ideation. This behavior is related to unbearable internal stress, thoughts, or mental pain, which NSSI assists in dismantling. To date, there is no generally approved therapy that assists in lowering NSSI. Ketamine is a sedative drug, presently at the focus of psychopharmacologic research, which was found to improve depression, when taken orally, and lower suicidal ideation, when given intravenously. Our aim is to assess the efficiency of intravenous ketamine in decreasing NSSI symptomology in women with a history of childhood sexual abuse presenting with such behavior. Participants will be recruited among hospitalized patients from the Tel-Aviv Medical Central psychiatric ward, who will present with either NSSI urges or behavior. The study design is a randomized control, double blind trial. Each patient will be assessed before, during, and after the trial by physical examination, blood tests and questionnaires. The patients will be randomized into research group (treated by ketamine and midazolam intravenously) or control group (treated intravenously via midazolam only). Our hypothesis is that treatment by intravenous ketamine will lower NSSI symptomology, and enable optimal treatment while being hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 y.o.
* Women
* Hospitalized
* Willing to sign the informed consent
* Fluent in Hebrew
* Reporting unbearable urge for self-injury and / or active NSSI behaviour) upon admittance, or on the preceding week.
* Not pregnant, nor breast feeding
* No history of drugs abuse
* No previous treatment with ketamine
* No psychotic disorder, nor severe physical condition (including unstable hypertension, arrhythmias or severe / active neurological condition)

Exclusion Criteria:

* Age < 18 year; Age >65 years
* Men
* Inability to sign informed consent, Non-Fluent in Hebrew.
* No report of NSSI, last NSSI event took place further than preceding week
* Active pregnancy or breast feeding
* History of drugs abuse
* Previous trial involving ketamine treatment during which no improvement was observed.
* Presence of psychotic disorder, and / or major physical condition (including unstable hypertension, arrhythmias or severe / active neurological condition).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-02-24 (Estimated); Study Completion 2024-02-24 (Estimated)

PRIMARY OUTCOMES:
Clinical measures - non suicidal self injuries symptoms | Four days prior to 1st treatment; after each intervention: 1 hour, 4 hours, 24 hours; next intervention will take place 3 days after (4 interventions altogether); 3 weeks post last intervention.
  Change in non suicidal self injuries symptoms will be measured by Brief Non-Suicidal Self-Injury Assessment (BNSSI), which assess the quality of self injuries (method of injury, time since last injury, causes of injury, motivation of self injury and bodily areas where injuries are most common).

SECONDARY OUTCOMES:
Clinical measures - biomarkers related to ketamine treatment - IL-6 | Four days prior to 1st treatment; 1 hour after 2nd intervention; 7 days later, 1 hour after 4th intervention; 3 weeks post last intervention.
  Changes in specific biomarkers as a result of ketamine treatment: interleukin 6 (IL-6).
Clinical measures - biomarkers related to ketamine treatment - hsCRP | Four days prior to 1st treatment; 1 hour after 2nd intervention; 7 days later, 1 hour after 4th intervention; 3 weeks post last intervention.
  Changes in specific biomarkers as a result of ketamine treatment: high sensitive C-Reactive Protein (hsCRP).
Clinical measures - biomarkers related to ketamine treatment - BDNF | Four days prior to 1st treatment; 1 hour after 2nd intervention; 7 days later, 1 hour after 4th intervention; 3 weeks post last intervention.
  Changes in specific biomarkers as a result of ketamine treatment - Brain Dendritic Neurotrophic Factor (BDNF).
Self reported questionnaires - depressive symptoms | BDI will be taken four days prior to 1st treatment; 1 hour after 2nd intervention; 7 days later, 1 hour after 4th intervention; 3 weeks post last intervention.
  Changes in depressive symptoms will be measured by Back Depression Inventory (BDI). Score scale from 1 to 40 points, higher score means more severe depression.
Self reported questionnaires - anxiety symptoms | DASS-21 will be taken four days prior to 1st treatment; 3 weeks post last intervention.
  Changes in anxiety symptoms will be measured by Depression, Anxiety and Stress Scale (DASS-21 Items).
  Score scale from 0 to 63 points, higher score means more severe anxiety symptoms.
Self reported questionnaires - Suicidal ideation | C-SSRS will be taken four days prior to 1st treatment.
  Changes in suicidal ideation will be measured by Columbia Suicide Severity Rating Scale (C-SSRS). This questionnaire assess severity of suicidal ideation, attempts and outcomes of attempted suicide.
Self reported questionnaires - Suicidal ideation | SSI will be taken four days prior to 1st treatment; 1 hour after 2nd intervention; 7 days later, 1 hour after 4th intervention; 3 weeks post last intervention.
  Changes in suicidal ideation will be measured by Scale for Suicidal Ideation (SSI). Score scale from 0 to 38 points, higher score means increased severity of suicidal ideation.
Self reported questionnaires - impulsivity | BIS-11 will be taken four days prior to 1st treatment four days; 3 weeks post last intervention.
  Changes in impulsive behavior will be measured by Barratt Impulsiveness Scale (BIS-11). This questionnaire assess impulsive behavior, with 30 items, including motor, attention and non-planning contributors. The factors are scored directly and reversibly, hence each factor assessed independently.
Self reported questionnaires - well being | WHO-5 will be taken four days prior to 1st treatment; 4 hour after 2nd intervention; 7 days later, 4 hour after 4th intervention; 3 weeks post last intervention.
  Patients well being will be measured by Well-Being Index (WHO 5). Higher score means greater well being.
Self reported questionnaires - Visual Analogue Scale (VAS) | VAS will be after each intervention: 1 hour, 4 hours, 24 hours; next intervention will take place 3 days after (4 interventions altogether).
  During the treatments, there will be an on going assessment by visual analogue scale, composed of items regarding symptomatology of non suicidal self-injuries, suicidality, Depression and anxiety.
Clinical measures - adverse effects | Adverse effects questionnaire will be taken after each intervention: 1 hour, 4 hours; next intervention will take place 3 days after (4 interventions altogether).
  During the treatments, the patient will be assessed for adverse effects of the infusion by ketamine side effects scale, including physical symptoms and psychotic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Miki Bloch, Prof., Principal Investigator — Tel Aviv University
Locations (1):
- Psychiatric Service, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No